CLINICAL TRIAL: NCT02143544
Title: Intra-aortic Balloon Counterpulsation in Patients Undergoing Cardiac Surgery: a Randomized Controlled Trial
Brief Title: Intra-aortic Balloon Counterpulsation in Patients Undergoing Cardiac Surgery
Acronym: IABCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, Professor of Cardiology, University of Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heart Institute
Record Dates: First submitted 2014-04-30; First posted 2014-05-21 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: Intra-aortic balloon counterpulsation; Cardiac surgery; High-risk patients
MeSH Terms: interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative intra-aortic balloon pump. (Active Comparator): Intervention: Preoperative placement of the intra-aortic balloon pump.
  Interventions: Device: Intra-aortic balloon pump.
- Control (No Intervention): No preoperative placement of the intra-aortic balloon pump.

INTERVENTIONS:
Device: Intra-aortic balloon pump. — Preoperative placement of the intra-aortic balloon pump.
  Arms: Preoperative intra-aortic balloon pump.

SUMMARY:
The hypothesis of the study is to evaluate if the preoperative placement of IABP reduces clinical complications in high-risk patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
High-risk patients undergoing cardiac surgery are at high risk for myocardial ischemia, arrhythmia, cardiogenic shock and other clinical complications. Different therapeutic options are available to support these patients in the perioperative period including inotropes, vasopressors, and vasodilators, and also assist devices such as intra-aortic balloon pump (IABP) and others.

IABP increases myocardial oxygen supply by increasing diastolic coronary perfusion pressure and decreases myocardial oxygen demand by reducing left ventricular afterload. Additionally, IABP can also improve cardiac output and systemic perfusion. The hypothesis of this randomized and controlled trial is that the placement of IABP immediately before the cardiac surgery reduces clinical complications in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or higher than 18 years old
* EuroSCORE equal to or higher than 6 or ejection fraction equal to or lower than 40%
* Written informed consent

Exclusion Criteria:

* Cardiogenic shock
* Acute myocardial infarction (AMI) < 48 hours
* Mechanical complications of AMI
* Peripheral vascular disease (aorta, iliac or femoral)
* Severe aortic regurgitation
* Neoplasm
* Pregnancy
* Tachyarrhythmia
* Procedures of the aorta
* Coagulopathy
* Thrombocytopenia
* Cardiac transplantation, congenital heart disease or endocarditis
* Refusal to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Composite 30-day mortality or major morbidity (mechanical ventilation > 24 hours, mediastinitis, surgical reexploration, stroke, cardiogenic shock, acute renal failure) | 30 days
  Composite outcome of 30-day mortality or incidence of patients presenting a major complication according to modified Society of Thoracic Surgeons (STS): mechanical ventilation > 24 hours, deep sternal wound infection/mediastinitis, surgical reexploration, stroke, cardiogenic shock and acute renal failure.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 30 days
  Number of days during mechanical ventilation.
IABP complications | 30 days
  Number of patients presenting one of the following: lower limb ischemia, mesenteric ischemia or bleeding.
Use of vasoactive agents | 30 days
  Number of days and dose of inotropes and vasopressors.
Evaluation of hemodynamic data | 48 hours
  Comparison of the following hemodynamic data between groups: heart rate, arterial pressure and cardiac output.
Levels of biomarkers | 7 days
  Comparison of the following biomarker levels between groups: pro-BNP (Brain natriuretic peptide), troponin I and Neutrophil gelatinase-associated lipocalin (NGAL), Heart-type Fatty Acid Binding Protein (H-FABP)
Echocardiographic parameters | 7 days
  Comparison of the following echocardiographic parameters between groups: left ventricular ejection fraction, cardiac output, left ventricular diastolic diameter, left ventricular systolic diameter and wall motion abnormalities.
30-day mortality | 30 days
  Death during hospital stay or death after hospital discharge until 30 days following the procedure
60-days mortality | 60 days
  Death until 60 days following the procedure
1-year mortality | 1 year
  Death until 1 year following the procedure
Costs | 30 days
  Comparison of overall costs between groups.
Acute Kidney Injury | 30 days
  Incidence of acute kidney injury according the Acute Kidney Injury Network (AKIN) classification.
Cardiovascular complications | 30 days
  Arrhythmias or myocardial ischemia within 30 days after randomization
Infectious complications | 30 days
  New infection or septic shock within 30 days after randomization
Delirium | 30 days
  Acute cognitive dysfunction diagnosed with the use of the CAM-ICU scale within 30 days after randomization
Bleeding | 24 hours
  Blood losses exceeding 100-300 mL per hour following ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Caldas JR, Panerai RB, Bor-Seng-Shu E, Ferreira GSR, Camara L, Passos RH, Salinet AM, Azevedo DS, de-Lima-Oliveira M, Galas FRBG, Fukushima JT, Nogueira R, Taccone FS, Landoni G, Almeida JP, Robinson TG, Hajjar LA. Intra-aortic balloon pump does not influence cerebral hemodynamics and neurological outcomes in high-risk cardiac patients undergoing cardiac surgery: an analysis of the IABCS trial. Ann Intensive Care. 2019 Nov 27;9(1):130. doi: 10.1186/s13613-019-0602-z. PMID 31773324
- [Derived] Caldas JR, Panerai RB, Bor-Seng-Shu E, Ferreira GSR, Camara L, Passos RH, de-Lima-Oliveira M, Galas FRBG, Almeida JP, Nogueira RC, Mian N, Gaiotto FA, Robinson TG, Hajjar LA. Dynamic cerebral autoregulation: A marker of post-operative delirium? Clin Neurophysiol. 2019 Jan;130(1):101-108. doi: 10.1016/j.clinph.2018.11.008. Epub 2018 Nov 22. PMID 30503909